CLINICAL TRIAL: NCT05014308
Title: Effect of Piezoelectric Alveolar Decortication on Post-Orthodontic Lower Incisors Stability: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Marwa Fahmy Saqat, master resident, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16011965
Record Dates: First submitted 2017-04-11; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Retention
Keywords: Retention; Relapse; Fibrotomy; Piezocision;
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- piezocision group (Experimental): piezocision surgical procedure was done according to Dibart's et al,
  Interventions: Procedure: Piezoelectric Alveolar Decortication, fibrotomy
- fiberotomy group (Experimental): the fiberotomy procedure followed Edward's et al
  Interventions: Procedure: Piezoelectric Alveolar Decortication, fibrotomy
- control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: Piezoelectric Alveolar Decortication, fibrotomy
  Arms: fiberotomy group; piezocision group

SUMMARY:
To assess the effect of piezocision on post-orthodontic lower anterior teeth stability as compared to fiberotomy and conventional Hawley retainers.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who had lower anterior irregularity (crowding, rotation, buccally or lingually displaced) will be selected.
2. Good oral hygiene, healthy gingiva and no evidence of bone loss as seen on the radiograph.
3. Healthy systemic conditions.
4. Patients pass the growth spurt according to cervical vertebral maturation method as described by Baccetti et al.
5. Availability of good quality records at pretreatment and post-treatment.

Exclusion Criteria:

1. Patients that has any signs of active periodontal disease or evidence of bone loss on the radiograph.
2. Patients with systemic disease such as osteoporosis and diabetes.
3. Smoking patients.
4. Study casts did not include all mandibular permanent incisors, canines, and first molars.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
lower incisors stability after 6 months | 6 months
  study models will be evaluated 6 months after debonding Incisor Irregularity Index of lower anterior teeth will be measured using a digital caliper
lower incisors stability after 12 months | 12 months
  study models will be evaluated 12 months after debonding Incisor Irregularity Index of lower anterior teeth will be measured using a digital caliper